CLINICAL TRIAL: NCT04955613
Title: 6Degrees VR System for Treatment of Phantom Limb Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: 6Degrees LTD (Industry)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202016500
Record Dates: First submitted 2021-05-05; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-05

CONDITIONS: Pain, Phantom
Keywords: phantom limb pain; VAS; Telerehabilitation
MeSH Terms: conditions — Phantom Limb | interventions — Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: A non-blinded controlled study of adults. Each patient admitted to the study will be randomly allocated to either the treatment or control group (provided standard care) in consecutive order.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Active Comparator): 12 sessions in total: sessions 1: Meeting with a doctor and physical therapist. sessions 2-11:Mirror therapy (standard care) for a total of 10 sessions over a period of 5 weeks (15-20 minutes per session).
  sessions 12: Meeting with a doctor and physical therapist.
  Interventions: Device: Mirror therapy
- MyMove/VR system (Active Comparator): sessions 1: Meeting with a doctor and physical therapist. sessions 2-11:MyMove devices and VR gear for a total of 10 sessions over a period of 5 weeks 15-20 minutes per session.
  sessions 12: Meeting with a doctor and physical therapist.
  Interventions: Device: MyMove/VR system

INTERVENTIONS:
Device: MyMove/VR system — The treatment system consists of two lightweight MyMove bands and Virtual-Reality (VR) gear. Proprietary software and content allow tracking of performance in real-time, with feedback to both the patient and treating - personnel.
  MyMove is a wearable device that allows patients with loss of upper limb function to operate computers, cellular phones, and similar devices. The technology is non-invasive and does not involve risk to the patient.
  Virtual-Reality (VR) gear is a wearable computer running within goggles that project content and allow for interaction using controllers.
  Arms: MyMove/VR system
Device: Mirror therapy — Mirror therapy or mirror visual feedback is a therapy for pain or disability that affects one side of the patient more than the other side
  Arms: Standard care

SUMMARY:
The treatment system consists of two light-weight MyMove bands and virtual-reality gear. Built-in software allows tracking of performance in real-time, with feedback to both the patient and treating personnel.

MyMove is a wearable device that allows patients with loss of upper-limb function to operate computers, cellular phones, and similar devices. The technology is non-invasive and does not involve risk to the patient.

MyMove+ is a Physical Medicine and Rehabilitation software intended for use in upper extremity and full-body conventional rehabilitation by:

1. Tracking motion and movement kinematics.
2. Guiding patients in the performance of physical exercises according to the treating practitioner's guidelines.

MyMove+ software is not intended for use in diagnosis, treatment or decision-making, or as a stand-alone device.

DETAILED DESCRIPTION:
A non-blinded controlled study of adults, ages 18-65, with unilateral, below-knee limb amputation.

All subjects will be initially evaluated by a single group of licensed physical- and occupational therapists. Following a structured introductory session, subjects will be assigned to MyMove devices and VR gear for a total of 10 sessions over a period of 5 weeks (15-20 minutes per session).

ELIGIBILITY:
Inclusion Criteria:

* Clearance by the treating physician.
* Unilateral below-knee amputation
* History of phantom-limb pain with an intensity of 5-or-greater (VAS scale)
* Pain is not responsive to conventional drugs or other standard treatment.
* Range of motion (knee) of 10-to-90 degrees.

Exclusion Criteria:

* Bilateral amputation
* History of phantom-limb pain with an intensity of 4-or-less (VAS scale)
* No prior attempt at therapy
* Declined by patient
* Pregnancy or other limitation related to special health-care groups.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2021-07-29 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Pain change | 12 months
  Demonstrate non-inferiority in comparison with existing treatments - change pain level by at least two visual analog scale (VAS) levels.
  VAS scale runs from 0 (pain-free) to 10 (extreme pain).

SECONDARY OUTCOMES:
Physical Rehabilitation Recovery | 12 months
  Demonstrate non-inferiority in comparison with existing treatments - change in range of motion over time.
  Angles measure from 0-120 degrees.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center', Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No
Data is system-specific to the MyMove bands and can only be analyzed with embedded algorithm reference.

REFERENCES:
- [Background] Hoffman HG, Boe DA, Rombokas E, Khadra C, LeMay S, Meyer WJ, Patterson S, Ballesteros A, Pitt SW. Virtual reality hand therapy: A new tool for nonopioid analgesia for acute procedural pain, hand rehabilitation, and VR embodiment therapy for phantom limb pain. J Hand Ther. 2020 Apr-Jun;33(2):254-262. doi: 10.1016/j.jht.2020.04.001. Epub 2020 May 30. PMID 32482376
- [Background] Ziegler-Graham K, MacKenzie EJ, Ephraim PL, Travison TG, Brookmeyer R. Estimating the prevalence of limb loss in the United States: 2005 to 2050. Arch Phys Med Rehabil. 2008 Mar;89(3):422-9. doi: 10.1016/j.apmr.2007.11.005. PMID 18295618
- [Background] Sherman RA, Sherman CJ, Parker L. Chronic phantom and stump pain among American veterans: results of a survey. Pain. 1984 Jan;18(1):83-95. doi: 10.1016/0304-3959(84)90128-3. PMID 6709380
- [Background] McCormick Z, Chang-Chien G, Marshall B, Huang M, Harden RN. Phantom limb pain: a systematic neuroanatomical-based review of pharmacologic treatment. Pain Med. 2014 Feb;15(2):292-305. doi: 10.1111/pme.12283. Epub 2013 Nov 13. PMID 24224475
- [Background] Ramachandran VS, Rogers-Ramachandran D. Synaesthesia in phantom limbs induced with mirrors. Proc Biol Sci. 1996 Apr 22;263(1369):377-86. doi: 10.1098/rspb.1996.0058. PMID 8637922
- [Background] Weeks SR, Anderson-Barnes VC, Tsao JW. Phantom limb pain: theories and therapies. Neurologist. 2010 Sep;16(5):277-86. doi: 10.1097/NRL.0b013e3181edf128. PMID 20827116